CLINICAL TRIAL: NCT05170620
Title: Research of Multiple Targeting CO2 Laser Ablation for the Treatment of Lower Anogenital Tracts' Precancerous Lesions
Brief Title: Research of Laser Ablation for the Treatment of Lower Anogenital Tracts' Precancerous Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20210134
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-01

CONDITIONS: Squamous Intraepithelial Lesions; Laser Burn
Keywords: laser; Cervical intraepithelial neoplasia; Vaginal intraepithelial neoplasia; Vulvar intraepithelial neoplasia; Anal intraepithelial neoplasia; Perianal intraepithelial neoplasia
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Uterine Cervical Dysplasia; Bowen's Disease | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients with squamous intraepithelial lesions of the lower anogenital tracts will receive laser ablation.
  Interventions: Procedure: laser ablation

INTERVENTIONS:
Procedure: laser ablation — Laser ablation will be done for the squamous intraepithelial lesions of the lower anogenital tracts.

SUMMARY:
Using multiple targeting CO2 laser ablation to treat the precancerous lesion of the female lower anogenital tracts and analyzing the data collected in the study, we aim to form the standard strategy of laser ablation method to increase the effective rate and lower the rate of relapse and progression.

DETAILED DESCRIPTION:
Patients diagnosed with CIN, VaIN, VIN, AIN or PAIN are recruited with exclusion of suspicion of malignant tumors. We use multiple targeting CO2 laser ablation to treat the precancerous lesion of the female lower anogenital tracts and then follow up the patients for at least two years. By analyzing the data collected in the study, we aim to form the standard strategy of laser ablation method to increase the effective rate and lower the rate of relapse and progression.

ELIGIBILITY:
Inclusion Criteria:

1. Had the history of sexual life.
2. Transferred to colposcopy examination and biopsy for abnormal screening of cervical cancer, contact bleeding of cervix, recurrent discomfort of vulva or abnormal signs of lower genital and anal tract. The pathology of biopsy indicate CIN, VaIN, VIN, AIN, or PaIN.
3. If CIN, the colposcopy manifests transformation zone-1 which means the lesion can totally be seen. However the consideration of fertility damage of resection overweighs the chance of suffering cancer.
4. The patients can accept multiple laser ablations and colposcopy examinations and follow-up at least 2 years.

Exclusion Criteria:

1. Patients who are suffering cancers of other systems and in treatment.
2. Patients suffering acute inflammation of lower genital and anal tracts.
3. The colposcopy and pathology examination suspect of cancer of lower genital and anal tract.
4. Patients suffering severe diseases such as insufficiency of liver and kidney function, diseases of blood system and other acute infections who will get heath harm from colposcopy and laser vaporization.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study focus on diseases of the female reproductive system.
Enrollment: 200 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological cure | up to at least two years
  No squamous intraepithelial lesions found by pathological examinations.

SECONDARY OUTCOMES:
HPV clearance | Every six months after initial treatment for at least two years
  The results of HPV tests are negative.

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Li, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No